CLINICAL TRIAL: NCT02001311
Title: Effect of Chlorhexidine Gel on Bacterial Count and Orthodontic Brackets During Fixed Orthodontic Treatment; In-vivo & In-vitro Study
Brief Title: Effect of Chlorhexidine Gel on Bacterial Count During Fixed Orthodontic Treatment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Dr. Samar Al-Bazi, Doctor, King Abdulaziz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 123
Record Dates: First submitted 2013-11-20; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Orthodontic Appliance Complication; Dental Caries
Keywords: chlorhexidine gel; orthodontic brackets; orthodontic patients; bacterial count; friction
MeSH Terms: conditions — Dental Caries | interventions — chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chlorhexidine gel (Experimental): anti microbial agent that prevents the formation of plaque and reduces caries risk
  Interventions: Drug: Chlorhexidine gluconate

INTERVENTIONS:
Drug: Chlorhexidine gluconate

SUMMARY:
This study investigates the benefit of using chlorhexidine gel as an antimicrobial agent in orthodontic patient to reduce caries risk and the possible consequential effect of this use on the orthodontic brackets used for the treatment.

The investigators hypothesis is that chlorhexidine gel use can reduce caries risk in orthodontic patients with out causing damage to the bonded ceramic or metal orthodontic brackets.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age range from 18-30 years.
* Fixed orthodontic treatment.
* All the patients are at the end of leveling and alignment stage.
* Initial bacterial count indicates high caries risk.
* All patients will be given good oral hygiene instruction at the first visit.
* The subjects had not taken antibiotics for at least 6 weeks before saliva sampling or during the experimental period.
* All subjects used a fluoride dentifrice twice a day.

Exclusion Criteria:

* Patients' age more or less then the age range specified.
* Removable orthodontic treatment.
* Patients at early stages of leveling and alignment.
* Initial bacterial count indicates low caries risk.
* Subjects that have taken antibiotics for at least 6 weeks before saliva sampling.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
mutants streptococcus count | 48 hours
  measures the change in bacterial count before and after application of the gel

SECONDARY OUTCOMES:
friction | 2 minutes
  measures static and dynamic friction in Newton

CONTACTS AND LOCATIONS:
Overall Officials: Samar M Al-Bazi, Principal Investigator — King Abdulaziz University

REFERENCES:
- [Derived] Al-Bazi SM, Abbassy MA, Bakry AS, Merdad LA, Hassan AH. Effects of chlorhexidine (gel) application on bacterial levels and orthodontic brackets during orthodontic treatment. J Oral Sci. 2016;58(1):35-42. doi: 10.2334/josnusd.58.35. PMID 27021538